CLINICAL TRIAL: NCT01067326
Title: The Effect of Tekturna on Endothelial Function and Endothelial Progenitor Cells in Patients With Early Atherosclerosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis ended all studies regarding Aliskiren.
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Novartis (Industry)
Responsible Party: Amir Lerman, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-007617; R01AG031750 (NIH); R01HL092954 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-11 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-01

CONDITIONS: Endothelial Dysfunction
Keywords: Endothelial Dysfunction; Endothelial Function; Tekturna; Endothelial Peripheral Arterial Tomography (EndoPAT); Progenitor Cells; renin inhibition; endothelial progenitor cells; early atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Active Comparator): 150 mg Aliskiren once daily for a period of 4 months.
  Interventions: Drug: Aliskiren
- Placebo (Placebo Comparator): 1 pill per day by mouth for 4 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — 150 mg Aliskiren once daily for a period of 4 months
  Other Names: Tekturna; Rasilez
  Arms: Aliskiren
Drug: Placebo — 1 pill per day by mouth for 4 months
  Arms: Placebo

SUMMARY:
We will study the hypothesis that long-term Tekturna treatment will improve endothelial function and the production and function of endothelial progenitor cells (EPCs) in patients with early atherosclerosis. Specifically, long-term Tekturna treatment will increase the Reactive Hyperemia Peripheral Arterial Tonometry indexes and increase the numbers and the function of circulating endothelial progenitor cells, compared to placebo, in association with a reduction in inflammation and oxidative stress.

DETAILED DESCRIPTION:
Aliskiren is a direct renin-inhibitor and may have beneficial effects on the vascular endothelium, similar to other antihypertensive therapies targeting the renin-angiotensin-aldosterone system (RAAS). The current study was designed to test the hypothesis that aliskiren improves endothelial function and increases the number of endothelial progenitor cells (EPCs) in normotensive patients with early atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. More than two of the following cardiovascular risk factors (determined by prescreen phone call): family history of cardiovascular disease, physical inactivity/sedentary lifestyle, obesity or overweight, family history of diabetes mellitus or hypertension, total cholesterol > 200 mg/dL, LDL > 130 mg/dL, HDL < 50 mg/dL, smoking, stress, or Triglycerides > 150 mg/dL
3. Demonstrated endothelial dysfunction (reactive hyperemia - EndoPAT score < 2.0) at time of screening

Exclusion Criteria:

1. Serum potassium > 5.0 mmol/L documented at any time prior to the study
2. History of any cardiovascular event (stroke, transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, coronary artery bypass grafting (CABG), percutaneous coronary intervention, hospitalization due to heart failure) during the 3 months prior to the study
3. Hypertension or hypotension (at Randomization): any patient with Mean Seated Systolic Blood Pressure (msSBP) ≥ 170 mmHg, msSBP < 100 mmHg or Mean Seated Diastolic Blood Pressure (msDBP) ≥ 110 mmHg
4. Congestive heart failure New York Heart Association (NYHA) class III and IV
5. Concomitant treatment with two (2) or more renin-angiotensin-aldosterone system blocking agents, e.g. Angiotensin Converting Enzyme Inhibitor (ACEI), Angiotensin II receptor blockers (ARB) or aldosterone-antagonist
6. Unstable serum creatinine
7. Second (II) or third (III) degree heart block without a pacemaker
8. Concurrent potentially life threatening arrhythmia or other uncontrolled arrhythmia
9. Clinically significant valvular heart disease
10. Known renal artery stenosis
11. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study drugs including, but not limited to, any of the following:

    * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
    * Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase
    * Evidence of hepatic disease as determined by a history of hepatic encephalopathy, a history of cirrhosis, esophageal varices, or a history of portocaval shunt
12. History of malignancy other than basal cell skin cancer within the past five years
13. Any concurrent life threatening condition with a life expectancy less than 2 years
14. History or evidence of drug or alcohol abuse within the last 12 months
15. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
16. History of hypersensitivity to any of the study drugs or to medications belonging to the same therapeutic class as the study drugs as well as known or suspected contraindications to the study drugs
17. History of noncompliance to medical regimens or unwillingness to comply with the study protocol
18. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
19. Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety
20. Persons directly involved in the execution of this protocol
21. Pregnant or nursing (lactating) women
22. Women of Child-Bearing Potential (WOCBP) unless postmenopausal for at least one year, surgically sterile or using effective methods of contraception as defined by local Health Authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Flammer AJ, Gossl M, Li J, Reriani M, Shonyo S, Loeffler D, Herrmann J, Lerman LO, Lerman A. Renin inhibition with aliskiren lowers circulating endothelial progenitor cells in patients with early atherosclerosis. J Hypertens. 2013 Mar;31(3):632-5. doi: 10.1097/HJH.0b013e32835c6d2d. No abstract available. PMID 23615219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Division of Cardiology at the Mayo Clinic in Rochester, Minnesota. 22 subjects were randomized to the study, 2 subjects were affected by the early study termination and thus have no follow-up data.
Period: Overall Study
Arm/Group | Aliskiren | Placebo
Started | 14 | 8
Completed | 12 | 5
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Early Study Termination | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aliskiren: 150 mg Aliskiren once daily for a period of 4 months. Not all baseline data were available from "started" subjects, therefore only baseline data for "completed" subjects is presented.
- Placebo: 1 pill per day by mouth for 4 months. Not all baseline data were available from "started" subjects, therefore only baseline data for "completed" subjects is presented.
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 12 | 5 | 17
Age Continuous [Mean (Standard Deviation); unit: years] — Not all baseline data were available from "started" subjects, therefore only baseline data for "completed" subjects is presented.
  years | 43.1 (17.5) | 51.0 (20.7) | 45.4 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Not all baseline data were available from "started" subjects, therefore baseline data for "completed" subjects is presented.
  Participants
    Female | 7 | 1 | 8
    Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants] — Not all baseline data were available from "started" subjects, therefore baseline data for "completed" subjects is presented.
  participants
    United States | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Progenitor Cells (EPC)
Description: Peripheral blood mononuclear cells were stained for EPC markers (cell-surface antigens CD34/CD133/KDR) and counted by flow-cytometry.
Time Frame: Baseline, 4 Months
Measure: Median (Inter-Quartile Range); unit: counts per 100,000 gated events
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 12 | 5
counts per 100,000 gated events
  Baseline | 24 [1 to 35] | 9 [3 to 19]
  4 Months | 3 [0 to 15] | 8 [2 to 11]
Statistical Analysis 1: Comparison: Aliskiren; Change in EPCs from baseline to 4 months; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

2. Secondary Outcome: Systolic Blood Pressure
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 12 | 5
mm Hg
  Baseline | 124.6 (12.2) | 118.8 (18.1)
  4 Months | 112.3 (12.4) | 116.2 (11.9)
Statistical Analysis 1: Comparison: Aliskiren; Difference in systolic blood pressure from baseline to 4 months; Test type: Superiority or Other; p = .006, t-test, 2 sided

3. Secondary Outcome: Diastolic Blood Pressure
Time Frame: Baseline, 4 Months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 12 | 5
mm Hg
  Baseline | 77.8 (9.9) | 68.6 (10.2)
  4 Months | 70.0 (11.6) | 67.6 (9.8)
Statistical Analysis 1: Comparison: Aliskiren; Difference in diastolic blood pressure from baseline to 4 months; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

4. Primary Outcome: Reactive Hyperemia Index (RHI)
Description: RHI was measured by the noninvasive endothelial peripheral arterial tomography (EndoPat) test. EndoPAT results are reported as the "Endoscore" (range 0-3); a score of 1.67 and lower indicates the need for immediate medical attention; a score between 1.68 and 2 indicates a need to reduce risk factors; a score above 2.1 indicates a healthy heart.
Time Frame: Baseline, 4 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 12 | 5
units on a scale
  Baseline | 1.93 [1.66 to 1.99] | 1.81 [1.63 to 2.05]
  4 Months | 1.73 [1.56 to 2.01] | 1.68 [1.41 to 2.19]
Statistical Analysis 1: Comparison: Aliskiren vs Placebo; P-value for intergroup comparison of change from baseline to month 4; Test type: Superiority or Other; p = 0.94, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: A study coordinator contacted the subjects by phone once weekly for the first month of the study and every month thereafter for the remainder of the study (4 months) to insure the safety of the subjects.
Arm/Group | Aliskiren | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5
Other Adverse Events (participants affected / at risk) | 0/12 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aliskiren (N=12) | Placebo (N=5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Irritated bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to safety concerns from the ALTITUDE trial; there was an unexpected increase in adverse events (non-fatal stroke, renal complications, hyperkalemia and hypotension). Novartis ended all studies regarding Aliskiren.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No